CLINICAL TRIAL: NCT00445575
Title: Effect of Risedronate on Bone Morbidity in Fibrous Dysplasia of Bone
Acronym: PROFIDYS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBM 03-54; AFSSAPS 060834
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Fibrous Dysplasia of Bone
Keywords: fibrous dysplasia of bone; Mac Cune Albright syndrome; bisphosphonates; risedronate
MeSH Terms: conditions — Fibrous Dysplasia of Bone | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): treatment duration: 1 year
  Interventions: Drug: risedronate
- 2 (Placebo Comparator): treatment duration: 1 year
  Interventions: Drug: placebo
- 3 (Experimental): duration treatment: 3 years
  Interventions: Drug: risedronate
- 4 (Placebo Comparator): treatment duration: 3 years
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: risedronate — During two months courses, every 6 months : 30mg tablet/day for adults and 10mg/day or 20mg/day for children, according to the age and weight of the child.
  Arms: 1
Drug: placebo — placebo and risedronate have exactly the same aspect. During two months courses, every 6 months : 30mg tablet/day for adults and 10mg/day or 20mg/day for children, according to the age and weight of the child.
  Arms: 2
Drug: risedronate — During two months courses, every 6 months : 30mg tablet/day for adults and 10mg/day or 20mg/day for children, according to the age and weight of the child.
  Arms: 3
Drug: placebo — placebo and risedronate have exactly the same aspect. During two months courses, every 6 months : 30mg tablet/day for adults and 10mg/day or 20mg/day for children, according to the age and weight of the child.
  Arms: 4

SUMMARY:
This trial is intended to test the efficacy of an oral bisphosphonate (risedronate) to decrease bone pain and improve radiological aspect in fibrous dysplasia of bone.

DETAILED DESCRIPTION:
In open pilot studies, it has been suggested that bisphosphonates may alleviate bone pain and help decrease the surface of osteolytic lesion in patients with fibrous dysplasia of bone (FD). So, in this randomized placebo controlled trial, we test the hypothesis that the bisphosphonate risedronate reduces bone pain in patients with FD (study I, one year duration) and decrease osteolytic lesions (study II, three years duration). Patients will take risedronate during 2 months courses, every 6 months or a matching placebo. Dosage will be : 30mg tablet/day for adults and 5mg tablet x 2,4 according to the age and weight of the child. All participants will receive calcium and vitamin D. All patients with renal phosphate wasting will receive an oral phosphate supplement.

ELIGIBILITY:
Inclusion Criteria:

* Study I: patients with FD, with bone pain intensity above 3 on visual analogical scale from 0 to 10
* Study II: patients with FD with at least one osteolytic lesion and no current bone pain

Exclusion Criteria:

* patients < 8 years old
* other diseases affecting bone metabolism
* patients with malignant diseases or other conditions likely to reduce their life expectancy to less than 3 years
* patients with history of significant upper gastrointestinal disorders
* renal failure (creatinine clearance < 25 ml/mn)
* severe liver disease
* history of iritis or uveitis
* rickets or osteomalacia
* allergy to bisphosphonates
* pregnancy or lactation
* prior treatment with a bisphosphonate
* laboratory abnormalities that may be considered as clinically significant by trial physicians

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-07-22 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Intensity of bone pain, assessed by visual analogical scale ranging from 0 to 10, on the most painful site. | one year
Surface of osteolytic lesions at three years. Radiological improvement. | Three years

SECONDARY OUTCOMES:
Variation of biochemical markers of bone turnover at three years | three years
Number of painful sites | one year
Improvement in quality of life | one to three years
Variation in bone mineral density of the femoral neck at three years | three years

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND D CHAPURLAT, MD PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; PHILIPPE ORCEL, MD PhD, Study Director — HOPITAL LARIBOISIERE; SOCRATES D PAPAPOULOS, MD PhD, Study Chair — Leiden University Medical Center
Locations (8):
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- France (3):
  - Hopital E Herriot, Lyon
  - Hopital Lariboisiere, Paris
  - Hopital Cochin, Paris
- Germany (3):
  - Hospital Benjamin Franklin, Berlin
  - Cologne Clinical Centre, Cologne
  - Heildeberg Clinical Centre, Heidelberg
- Leids Universitair Medisch Centrum, Leiden, Netherlands

REFERENCES:
- See also: Related Info — http://www.dysplasie-fibreuse-des-os.info/fr/accueil.html